CLINICAL TRIAL: NCT03768908
Title: A Multicentre Randomised Comparative Clinical Trial of the Efficacy of Artesunate + Amodiaquine Versus Artemether-lumefantrine (Coartem®) for the Treatment of Uncomplicated Childhood Plasmodium Falciparum Malaria in Zanzibar
Brief Title: Efficacy of Artesunate + Amodiaquine Versus Artemether-lumefantrine for Falciparum Malaria in Zanzibar, 2005
Acronym: ACOII
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Professor Anders Björkman (Other)
Collaborators: Zanzibar Malaria Control Programme (Other Government)
Responsible Party: Sponsor-Investigator, Professor Anders Björkman, Professor, Karolinska Institutet
Organization: Karolinska Institutet (Other)
Allocation: Randomized | Masking: None | Purpose: Treatment
Other Study IDs: ACO II
Record Dates: First submitted 2018-12-03; First posted 2018-12-07 (Actual); Last update posted 2018-12-07 (Actual); Status verified 2018-12

CONDITIONS: Plasmodium Falciparum Malaria
Keywords: Artemether-Lumefantrine; Coartem; Artesunate; Amodiaquine; Zanzibar
MeSH Terms: conditions — Malaria, Falciparum | interventions — Artemether, Lumefantrine Drug Combination; amodiaquine, artesunate drug combination

STUDY DESIGN:
Intervention Model Description: A multicentre randomised comparative clinical trial of the efficacy of ASAQ versus AL for the treatment of uncomplicated childhood Plasmodium falciparum malaria.
Masking Description: No blinding was done due to the different drug formulations and regimens.
Oversight: Data Monitoring Committee: No

ARMS (2):
- Treatment with artesunate + amodiaquine (Active Comparator): Co-administration of a daily dose of artesunate (Arsumax) 4mg/kg and amodiaquine (Flavoquine) 10mg/kg for 3 days, under direct observation. Children <12months <10kg: artesunate (Arsumax) 50mg - 0.5tab/day + amodiaquine (Flavoquine) 153mg - 0.5tab/day; Children 12-59months 10-20kg: artesunate (Arsumax) 50mg - 1 tab/day + amodiaquine (Flavoquine) 153mg 1 tab/day.
  Interventions: Drug: Artesunate + Amodiaquine
- Treatment with artemether-lumefantrine (Coartem®) (Active Comparator): Artemether-lumefantrine (Coartem®) - artemether 1.3mg/kg + lumefantrine 4mg/kg administered twice daily, both doses under direct observation either in the clinic or in the patient's home. Children <60 months, 5-14kg: 1 tab/dose; Children <60 months >14kg: 2 tabs/dose.
  Interventions: Drug: Artemether-lumefantrine

INTERVENTIONS:
Drug: Artemether-lumefantrine — Three day treatment with Artemether-lumefantrine, 2 doses a day under direct observation
  Other Names: Coartem®
  Arms: Treatment with artemether-lumefantrine (Coartem®)
Drug: Artesunate + Amodiaquine — Three day treatment with Artesunate + Amodiaquine, co-administered, a dose a day under direct observation
  Other Names: ASAQ
  Arms: Treatment with artesunate + amodiaquine

SUMMARY:
The primary objective of the study was to determine the PCR-APCR up to day 42 in children <60 months of age, weighing ≥5kg with uncomplicated malaria, treated with either artesunate+ amodiaquine (ASAQ) or artemether-lumefantrine (AL; Coartem®).

Secondary objectives included: clinical and laboratory assessment of drug tolerability and safety, evaluation of possible correlation between drug bioavailability and clinical outcome, comparison of efficacy data with the pre-implementation "ACO I" study, parasite and fever clearance, gametocyte carriage, and possible selection of mutations related to quinoline resistance.

DETAILED DESCRIPTION:
All children in the right age group presenting with clinical signs of malaria at the study site were considered possible study subjects. The guardians of these children were informed about the study orally in Swahili according to the informed consent form. Those who were not willing to participate in the study were treated according to local standard procedure.

On day 0 the patient was tested for parasites using light microscopy on Giemsa stained blood films. A detailed clinical history and a clinical examination including an axillary temperature was assessed. Haemoglobin was assessed and blood samples were collected on filter paper for each child for genotyping of the parasites as well as for possible determination of blood levels of different antimalarial drugs.

The guardian was asked to bring their child back to the study site on day 1, 2, 3, 7, 14, 21, 28, 35 and 42. If they failed to do so they were visited in their homes to assure proper follow-up. At each follow-up the investigator asked about concomitant medication and adverse events, carefully filling out the clinical report form (CRF).

If, during the follow-up between day 14 and 42, a child previously enrolled in the study presented with fever, all tests and examinations were run as on day 0. If the child was clinically and parasitologically diagnosed with malaria again, he was treated as a new infection. If diagnosed with severe malaria during the follow-up period the patient was given rescue treatment (oral or intravenous Quinine) and withdrawn from the study. Each time an enrolled child presented at the site the CRF was completed with regards to clinical and laboratory status, treatment given and possible adverse events.

Clinical and laboratory assessments included:

Malaria smear: Giemsa stained thick blood films examined using electrical or sunlight microscope at the study site by an experienced microscopist. The number of parasites were calculated as the number of parasites seen against 200 leucocytes in the thick blood film and recorded in the CRF for the correct occasion. The slides were stored for quality controls double-check (10% of all slides) centrally.

Haemoglobin: Haemoglobin levels were measured by the HaemoCue™ method using blood samples collected on cuvettes. The Hb levels were recorded in the CRF for each occasion.

Full Blood Picture (FBP) and Liver Function Test (LFT): FBP and LFT were performed in the Kivunge Study Site sub-population only (GLP Sub Study). FBP was obtained using the Cell-Dyn 1700™ Haematology Analyser (Abbott Laboratories, USA). LFT, including ALT, AST, Gamma-GT, albumin and bilirubin, was obtained using the BTS-310™ Photometer UV-VIS (BioSystems, Spain).

Temperature and Clinical history: A medical doctor/officer measured the patient's axillary temperature using an electronic thermometer and took a detailed clinical history as well as performed a clinical examination.

PCR Filter paper sample: Blood samples were collected on Whatman FTA filter papers. When dry, each filter paper sample was stored in separate plastic bags at -20ºC (Kivunge) or +4ºC (Micheweni) until regularly transferred to Kivunge for -20ºC long term storage.

HPLC samples (Kivunge only): Approximately 5ml of venous blood was drawn from each patient on days 0 and 7 for FBP and LFT tests. In the ASAQ group 100 µl of this blood was collected on special filter papers for high pressure liquid chromatography (HPLC) analysis of amodiaquine levels. In the AL group 100 µl of plasma (separated by centrifugation at >3000rpm for 10min) was collected on special filter papers for HPLC analysis of lumefantrine levels. All remaining (minimum 2ml) of plasma was collected and kept at -20ºC as a back-up.

Molecular analyses: PCR genotyping of merozoite surface protein 2 (msp2), considered the most informative single genetic marker for multiplicity of P. falciparum infections, was performed to differentiate reinfections from true recrudescence. Paired PCR results were compared between day 0 and at the time of recurrent parasitaemia from day 14 up to day 42. The outer conserved region of the polymorphic repetitive block 3 of msp2 was amplified in an initial reaction followed by two nested reactions with oligonucleotide primers specific for the two allelic families FC27 and IC/3D7, using a standard protocol. The pfmdr1 Y86N and pfcrt K76T genes' Single Nucleotide Proteins (SNPs) analysis was done according to established AluI restriction-based PCR-RFLP protocols. All molecular analyses were performed at the Malaria Research Unit, KI, Sweden.

ELIGIBILITY:
Inclusion Criteria:

* Weight ≥5kg
* No general danger signs or severe malaria present (see 4.4.2.1 & 4.4.2.2)
* History of fever within 24 hours OR axillary temperature ≥ 37.5Cº
* No other cause of fever is detectable
* No severe malnutrition
* Patient has parasite counts between 2000-200,000/ul (50-5000/200 white blood cells)
* Guardian/Patient has understood the procedures of the study and is willing to participate
* Patient able to come for stipulated follow up visits and has easy access to the Study Site

Exclusion Criteria:

General Danger Signs and Complications:

* Not able to drink or breastfeed
* Vomiting everything
* Recent history of convulsions
* Lethargic or unconscious
* Unable to sit or stand (as appropriate for age)
* History of allergy to test drugs
* History of intake of any drugs other than paracetamol and aspirin within 3 days

Signs of Severe Malaria:

* Altered consciousness
* Repeated convulsions
* Inability of oral intake
* Severe anaemia (Hb <5gm/dl)
* Difficulty in breathing (pulmonary oedema, Respiratory Distress Syndrome)
* Shock (small pulse, cold extremities)
* Hypoglycaemia
* Haemoglobinuria (dark coloured urine or Coca-Cola urine)
* Kidney failure (little or no urine in a well-hydrated patient)
* Jaundice (yellow colouring of eyes)
* Hyperpyrexia (temperature above 39.5ºC) in combination with other signs
* Hyperparasitaemia (more than 5% red blood cells parasitized or >200,000 parasites/µl)
* Spontaneous bleeding (Disseminated Intravascular Coagulation)

Max Age: 60 Months | Sex: All
Age Groups: Child
Enrollment: 359 (Actual)
Dates: Start 2005-01-05 (Actual); Primary Completion 2005-07-11 (Actual); Study Completion 2005-07-11 (Actual)

PRIMARY OUTCOMES:
PCR adjusted parasitological cure rates by day 42 | 42 days
  Comparing PCR adjusted parasitological cure rate (PCR-APCR) between the two treatment options up to day 42. Parasitological cure will be adjusted using PCR genotyping of msp2 marker. Recrudescence is defined as the presence of at least one matching allelic band, and reinfection as the absence of any matching allelic band on day 0 and day of recurring parasitaemia. Patients with recurrent parasitaemia having missing filter paper sample or negative PCR results will be considered uncertain with regards to PCR adjusted outcome.

SECONDARY OUTCOMES:
The clinical and parasitological response outcome (i.e. cure rates) on days 14, day 28 and 42. | 42 days
  Comparing proportion of response outcomes according to standard WHO classification i.e., cure rates on days 14, day 28 and 42. Defined as the absence of both re-parasitaemia and clinical symptoms suggestive of severe malaria during follow-up to the respective days.

OTHER OUTCOMES:
Clinical and laboratory assessment of drug tolerability and safety i.e., incidence of adverse events. | 42 days
  Proportion of patients reporting any adverse event (AE) in the two study arms. The intensity of an adverse event was determined according to the following definitions: mild, moderate, severe, unknown. AEs were be categorized according to if there is a likely causal relationship between the event and the medical products: probably, possibly, unlikely.
Fever clearance in the two study arms | 42 days
  Fever clearance was determined by a medical doctor/officer who measured the patient's axillary temperature using an electronic thermometer and took a detailed clinical history as well as performed a clinical examination. All details were recorded in the CRF.
Parasite clearance and gametocyte carriage in the two study arms | 42 days
  Clearance of parasites and gametocyte carriage were determined by Giemsa stained thick blood films were examined using electrical or sunlight microscope at the study site by an experienced microscopist. The number of parasites were calculated as the number of parasites seen against 200 leucocytes in the thick blood film and recorded in the CRF for the correct occasion. The slides were stored for quality controls, 10% of all slides were double-checked centrally.
Proportion of mutations related to Quinoline resistance at day0 and day of recurrent infection in the two study arms | 42 days
  Proportions of single nucleotide polymorphisms at pfmdr1 Y86N and pfcrt K76T determined by established AluI restriction-based PCR-RFLP.

CONTACTS AND LOCATIONS:
Overall Officials: Johan Stromberg, Principal Investigator — Karolinska Institutet; Mwinyi I Msellem — Zanzibar Malaria Control Programme; Andreas Martensson — Karolinska Institutet

REFERENCES:
- [Background] Holmgren G, Hamrin J, Svard J, Martensson A, Gil JP, Bjorkman A. Selection of pfmdr1 mutations after amodiaquine monotherapy and amodiaquine plus artemisinin combination therapy in East Africa. Infect Genet Evol. 2007 Sep;7(5):562-9. doi: 10.1016/j.meegid.2007.03.005. Epub 2007 Mar 31. PMID 17467344